CLINICAL TRIAL: NCT02396849
Title: Modulation Of Airway Reactivity With Chronic Mechanical Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Tepper, Robert Tepper, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4689673; 5R01HL048522 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) (Experimental): Use of a CPAP machine for at least 5 days per week for 28 days
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Continuous Positive Airway Pressure (CPAP) Sham (Sham Comparator): Use of a sham CPAP machine for at least 5 days per week for 28 days
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) Sham

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Subjects assigned to this group will be asked to use the CPAP machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
  Arms: Continuous Positive Airway Pressure (CPAP)
Device: Continuous Positive Airway Pressure (CPAP) Sham — Subjects assigned to this group will be asked to use the CPAP Sham machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
  Arms: Continuous Positive Airway Pressure (CPAP) Sham

SUMMARY:
The purpose of this study is to see if the use of a machine called CPAP will help children with asthma breathe better. CPAP is a machine that produces airflow to help people with breathing problems. To use it, you will wear a mask connected by a hose to the CPAP machine. We believe that use of CPAP may be a treatment for children with asthma.

DETAILED DESCRIPTION:
During the previous funding period of this project, our laboratory demonstrated that chronic mechanical strain imposed on the airways in vivo using continuous positive airway pressure (CPAP) results in a dramatic reduction in airway reactivity in vivo in mice, ferrets and rabbits1-3. Lungs, airways and airway smooth muscle (ASM) tissues isolated from CPAP-treated animals studied in vitro exhibited lower responsiveness to bronchoconstrictors1-3. We also observed this suppression of airway responsiveness by chronic mechanical strain in a rabbit model of allergic asthma5. These animal studies led to a small clinical trial in which adults with asthma were treated with nocturnal CPAP for 1 week. CPAP caused a significant reduction in airway reactivity in these patients6. This novel approach for treating airway hyper-reactivity is currently being evaluated in a NIH multi-center Phase II clinical trial of adults with mild to moderate asthma (U01 HL108730).

ELIGIBILITY:
Inclusion Criteria:

* Children 8-17 yrs olds with severe asthma (N=120) will be recruited from the Pediatric High Risk Asthma Clinic and Pulmonary Clinics at Riley Hospital for Children at Indiana University Health.
* Severe asthma will be defined by the need for medication therapies following steps 4-6 according to the National Institutes of Health's Asthma Care Quick Reference, September 2012 or high dose of inhaled corticosteroids
* On a stable regimen of asthma medications for at least 8 weeks prior to enrollment without systemic corticosteroids for ≥ 4 weeks

Exclusion Criteria:

* Obese (>95% predicted BMI)
* Congenital heart disease or chronic lung disease
* History of pneumothorax
* Inability to perform pulmonary function testing
* Oxygen saturation <93%
* forced expiratory volume at one second (FEV1) <70% predicted
* Provocative concentration causing a 20% drop in FEV1 from baseline (PC20) ≥16 mg/ml of methacholine.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tepper, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Praca E, Jalou H, Krupp N, Delecaris A, Hatch J, Slaven J, Gunst SJ, Tepper RS. Effect of CPAP on airway reactivity and airway inflammation in children with moderate-severe asthma. Respirology. 2019 Apr;24(4):338-344. doi: 10.1111/resp.13441. Epub 2018 Nov 16. PMID 30444283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 were excluded based on screening criteria, two subjects (one in each group) were lost to follow-up, two (one in each group) did not tolerate the equipment and two (one in each group) did not undergo Methacholine challenge at V2 due to the presence of asthma symptoms.
Groups:
- Continuous Positive Airway Pressure (CPAP): Use of a CPAP machine for at least 5 days per week for 28 days
  CPAP: Subjects assigned to this group will be asked to use the CPAP machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
- Continuous Positive Airway Pressure (CPAP) Sham: Use of a sham CPAP machine for at least 5 days per week for 28 days
  CPAP Sham: Subjects assigned to this group will be asked to use the CPAP SHAM machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Continuous Positive Airway Pressure (CPAP) Sham
Started | 29 | 30
Completed | 27 | 28
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Did not tolerate intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- CPAP: Use of a CPAP machine for at least 5 days per week for 28 days
  CPAP: Subjects assigned to this group will be asked to use the CPAP machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
- CPAP Sham: Use of a sham CPAP machine for at least 5 days per week for 28 days
  CPAP Sham: Subjects assigned to this group will be asked to use the CPAP SHAM machine for a minimum of 4 hours/night at least 5 days/week for a total of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | CPAP | CPAP Sham | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (2.5) | 11.7 (2.5) | 11.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 16 | 16 | 32
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 28 | 55
Methacholine Bronchial Challenge [Mean (Standard Deviation); unit: mg/mL] — Methacholine bronchial challenge was performed using the 5-breath protocol (DeVilbiss646 with KoKo dosimeter: 9 μL/breath) with quadrupling concentrations starting with 0.0625 mg/mL and continuing until forced expiratory volume at one second (FEV1) decreased by 20% or Methacholine concentration of 16 mg/mL was inhaled.
  mg/mL | 2.9 (4.5) | 3.2 (4.3) | 3.09 (4.38)

OUTCOME MEASURES:

1. Primary Outcome: Change in Airway Reactivity From Baseline (Visit 1) and 4 Weeks (Visit 2)
Description: The change in airway reactivity measured prior to and after 4 weeks of either CPAP or SHAM treatment. Methacholine bronchial challenge was performed using the 5-breath protocol (DeVilbiss646 with KoKo dosimeter: 9 μL/breath) with quadrupling concentrations starting with 0.0625 mg/mL and continuing until FEV1 decreased by 20% (PC20) or Methacholine concentration of 16 mg/mL was inhaled.
Time Frame: baseline (visit 1) and 4 weeks (visit 2)
Population: One subject in each group did not undergo Methacholine challenge at V2 due to the presence of asthma symptoms
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | CPAP | CPAP Sham
Number analyzed (Participants) | 26 | 27
mg/mL
  Visit 1 | 3.0 (4.6) | 3.2 (4.4)
  Visit 2 | 5.3 (8.9) | 4.3 (6.8)

2. Secondary Outcome: Change in Airway Inflammation From Baseline (Visit 1) and 4 Weeks (Visit 2)
Description: Airway Inflammation assessed as the change in the percentage eosinophils in the induced sputum measured prior to and after 4 weeks of Continuous Positive Airway Pressure (CPAP) or sham CPAP treatment.
Time Frame: baseline (visit 1) and 4 weeks (visit 2)
Population: The overall success rate in obtaining quality sputum samples was 57%; however, only 10 CPAP and 12 sham subjects had quality samples at both study visits.
Measure: Mean (Standard Deviation); unit: Percentage of sputum eosinophils
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Continuous Positive Airway Pressure (CPAP) Sham
Number analyzed (Participants) | 10 | 12
Percentage of sputum eosinophils
  Study Visit 1 | 6.2 (10.1) | 3.9 (5.0)
  Study Visit 2 | 3.6 (6.4) | 5.4 (8.2)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse event were described as an asthma exacerbation requiring oral corticosteroids during the study period.
Arm/Group | CPAP | CPAP Sham
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 5/29 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPAP (N=29) | CPAP Sham (N=30)
asthma exacerbation treated with oral corticosteroids (Respiratory, thoracic and mediastinal disorders) | 5 | 3

LIMITATIONS AND CAVEATS:
We evaluated only children with moderate-severe asthma, the results cannot be extrapolated to children with mild or moderate asthma. A major limitation of our study was the limited number of subjects we could recruit from a single pediatric center. Our evaluation of airway inflammation was limited to induced sputum rather than bronchoalveolar lavage, which would not have been an acceptable risk in our children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT02396849/Prot_SAP_000.pdf